CLINICAL TRIAL: NCT02367040
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Copanlisib in Combination With Rituximab in Patients With Relapsed Indolent B-cell Non-Hodgkin's Lymphoma (iNHL) - CHRONOS-3
Brief Title: Copanlisib and Rituximab in Relapsed Indolent B-cell Non-Hodgkin's Lymphoma (iNHL)
Acronym: CHRONOS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17067; 2013-003893-29 (EudraCT Number)
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma,Non-Hodgkin
Keywords: Clinical trial, Phase III; Phosphatidylinositol-3-kinase; Non-Hodgkin's lymphoma; Indolent B-cell non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Copanlisib + Rituximab (Experimental): Combination of the Copanlisib and rituximab
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946); Drug: Rituximab
- Placebo + Rituximab (Placebo Comparator): Combination of Copanlisib placebo and rituximab
  Interventions: Drug: Placebo; Drug: Rituximab

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — Copanlisib is supplied as lyophilized preparation in a 6 mL injection vial. The total amount of copanlisib per vial is 60 mg. The solution for IV infusions is obtained after reconstitution with normal saline solution. Dosing will be administered on Days 1, 8 and 15 of each 28-day cycle. Copanlisib will be administered before rituximab.
  Arms: Copanlisib + Rituximab
Drug: Placebo — Placebo is supplied as lyophilized preparation in a 6 mL injection vial. The developed placebo lyophilisate is equivalent to the 60 mg copanlisib formulation, with regard to the composition of excipients and the instructions for reconstitution and dose preparation. Placebo dosing will be administered on Days 1, 8 and 15 of each 28-day cycle. Placebo will be administered before rituximab.
  Arms: Placebo + Rituximab
Drug: Rituximab — Rituximab dose 375 mg/m2 body surface weekly during Cycle 1 on Days 1, 8, 15 and 22, and then on Day 1 of Cycles 3, 5, 7 and 9.The solution for IV infusions is obtained after reconstitution of a calculated concentration of 1 to 4 mg/ml rituximab into an infusion bag containing sterile, pyrogen-free sodium chloride 9 mg/ml (0.9%) solution for injection or 5% D-Glucose in water.

SUMMARY:
The purpose of this study was to evaluate whether copanlisib in combination with rituximab is superior to placebo in combination with rituximab in prolonging progression free survival (PFS) in patients with relapsed iNHL who have received one or more lines of treatment, including rituximab and who either had a treatment-free interval of ≥ 12 months after completion of the last rituximab-containing treatment, or who are unwilling to receive chemotherapy/for whom chemotherapy is contraindicated on reason of age, comorbidities, and/or residual toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Indolent non-Hodgkin's lymphoma (iNHL) in CD20 positive patients, with histological subtype limited to:

  * Follicular lymphoma(FL) grade1-2-3a
  * Small lymphocytic lymphoma(SLL) with absolute lymphocyte count <5x10*9/L at study entry
  * Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM)
  * Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)
* Patients must have relapsed (recurrence after complete response or presented progression after partial response) after the last rituximab-, rituximab biosimilars-, or anti-CD20 monoclonal antibody (e.g. obinutuzumab)-containing therapy (other previous treatment lines after rituximab are allowed). A previous regimen is defined as one of the following: at least 2 months of single-agent therapy (less than 2 months of therapy is allowed for patients who responded to single-agent rituximab, rituximab biosimilars, or anti-CD20 monoclonal antibody); at least 2 consecutive cycles of polychemotherapy; autologous transplant; radioimmunotherapy. Previous exposure to PI3K is acceptable (except to copanlisib) provided there is no resistance. Patients with prior intolerance to PI3K inhibitors other than copanlisib are eligible.
* Non-WM must have at least one bi-dimensionally measurable lesion (which has not been previously irradiated) according to the Lugano Classification. For patients with splenic MZL (Marginal-zone lymphoma) this requirement may be restricted to splenomegaly alone since that is usually the only manifestation of measurable disease.
* Patients affected by WM who do not have at least one bi-dimensionally measurable lesion in the baseline radiologic assessment must have measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level ≥ 2 x upper limit of normal (ULN) and positive immunofixation test .
* Male or female patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of at least 3 months
* Availability of fresh tumor tissue and/or archival tumor tissue for central pathology(obtained within 5 years of the consent date) at Screening
* Adequate baseline laboratory values collected no more than 7 days before starting study treatment
* Left ventricular ejection fraction ≥ 45%
* Patients must either:

  * have had a progression-free and treatment-free interval of at least 12 months after completion of the rituximab-, rituximab biosimilars-, or anti-CD20 monoclonal antibody-containing treatment OR
  * be considered unfit to receive chemotherapy on reason of age, concomitant morbidities, and/or residual toxicity from previous treatments, or unwillingness to receive chemotherapy. These patients must also have had a progression-free and treatment-free interval of at least 6 months after completion of the last rituximab-, rituximab biosimilars-, or anti-CD20 monoclonal antibody-containing treatment. Patients in whom chemotherapy is contraindicated are defined by one of the following features:

    * Age ≥ 80 years
    * Age < 80 years and at least 1 of the following conditions:

      * at least 3 grade 3 CIRS-G comorbidities OR
      * at least 1 grade 4 CIRS-G comorbidity (if compatible to participation in the study).

Exclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma grade 3b or transformed disease, or chronic lymphocytic leukemia
* Progression free interval or treatment free interval of less than 12 months since the last rituximab-, rituximab biosimilars-, or anti-CD20 monoclonal antibody (e.g. obinutuzumab)-containing treatment(including maintenance with these drugs). For patients considered unwilling/unfit to receive chemotherapy : progression free interval or treatment free interval of less than 6 months since the last rituximab-, rituximab biosimilars-, or anti-CD20 monoclonal antibody-containing treatment (including maintenance with these drugs), as assessed by the investigator
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* Known lymphomatous involvement of the central nervous system
* Patients with HbA1c > 8.5% at Screening
* Known history of human immunodeficiency virus (HIV) infection
* Hepatitis B (HBV) or hepatitis C (HCV). Patients positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti- HCV antibody will be eligible if they are negative for HCV-RNA
* Documented evidence of resistance to prior treatment with idelalisib or other PI3K inhibitors.
* Prior treatment with copanlisib
* Cytomegalovirus (CMV) infection. Patients who are CMV PCR positive at baseline will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (160):
- United States (16):
  - West Covina, California
  - Ashland, Kentucky
  - Louisville, Kentucky
  - Bethesda, Maryland
  - Las Vegas, Nevada
  - Montvale, New Jersey
  - MSK Basking Ridge, New Jersey, New Jersey
  - MSK Bergen, New Jersey, New Jersey
  - MSK Monmoth, New Jersey, New Jersey
  - MSK Westchester, Harrison, New York
  - MSK Commack, Long Island City, New York
  - MSK Rockville Centre, Long Island City, New York
  - New York, New York
  - Canton, Ohio
  - Salt Lake City, Utah
  - Spokane, Washington
- Argentina (4):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Córdoba
- Australia (2):
  - Ballarat, Victoria
  - Nedlands
- Austria (2):
  - Graz, Styria
  - Vienna
- Ottignies, Belgium
- Brazil (6):
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Barretos/SP, São Paulo
  - Jaú, São Paulo
  - São Paulo, São Paulo
  - São Paulo
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Temuco, Región de la Araucanía, Chile
- China (15):
  - Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shengyang, Liaoning
  - Chengdu, Sichuan
  - Ürümqi, Xinjiang
  - Hangzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Colombia (4):
  - Medellín, Antioquia
  - Bogota, Cundinamarca
  - Montería, Departamento de Córdoba
  - Cali, Valle del Cauca Department
- France (7):
  - Bayonne
  - Brest
  - Metz
  - Nice
  - Pessac
  - Poitiers
  - Saint-Herblain
- Germany (5):
  - München, Bavaria
  - Recklinghausen, North Rhine-Westphalia
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Berlin
- Greece (3):
  - Athens
  - Chaïdári
  - Pátrai
- Hong Kong (2):
  - Chai Wan
  - Hong Kong
- Hungary (5):
  - Budapest
  - Győr
  - Kaposvár
  - Pécs
  - Tatabánya
- Ireland (2):
  - Dublin
  - Galway
- Italy (4):
  - Udine, Friuli Venezia Giulia
  - Genoa, Liguria
  - Milan, Lombardy
  - Florence, Tuscany
- Japan (16):
  - Nagoya, Aichi-ken
  - Maebashi, Gunma
  - Kobe, Hyōgo
  - Nankoku, Kochi
  - Sendai, Miyagi
  - Ōmura, Nagasaki
  - Kurashiki, Okayama-ken
  - Hirakata, Osaka
  - Izumo, Shimane
  - Chuo-ku, Tokyo
  - Aomori
  - Fukuoka
  - Kumamoto
  - Niigata
  - Osaka
  - Yamagata
- Kaunas, Lithuania
- Malaysia (6):
  - Cheras
  - Kota Kinabalu
  - Kuala Lumpur
  - Kuala Selangor
  - Perak
  - Pulau Pinang
- Mexico (2):
  - Morelia, Michoacán
  - Monterrey, Nuevo León
- Tauranga, New Zealand
- Philippines (2):
  - City of Taguig
  - Pasig
- Poland (4):
  - Gdansk
  - Gdynia
  - Krakow
  - Lublin
- Porto, Portugal
- Romania (5):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Târgu Mureş
- Russia (9):
  - Chelyabinsk
  - Irkutsk
  - Kazan'
  - Kemerovo
  - Kirov
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Volgograd
- Singapore, Singapore
- Poprad, Slovakia
- South Africa (2):
  - George, Eastern Cape
  - Johannesburg, Gauteng
- South Korea (4):
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Hwasun Gun
  - Seoul
- Spain (5):
  - Majadahonda, Madrid
  - Málaga, Málaga
  - Barcelona
  - Madrid
  - Salamanca
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taipei
- Thailand (2):
  - Chiang Mai
  - Pathum Thani
- Turkey (Türkiye) (5):
  - Ankara
  - Istanbul
  - Izmir
  - Kayseri
  - Trabzon
- Ukraine (5):
  - Cherkasy
  - Dnipro
  - Kyiv
  - Lviv
  - Vinnitsa
- Vietnam (2):
  - Hà Nội
  - Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Matasar MJ, Capra M, Ozcan M, Lv F, Li W, Yanez E, Sapunarova K, Lin T, Jin J, Jurczak W, Hamed A, Wang MC, Baker R, Bondarenko I, Zhang Q, Feng J, Geissler K, Lazaroiu M, Saydam G, Szomor A, Bouabdallah K, Galiulin R, Uchida T, Soler LM, Cao A, Hiemeyer F, Mehra A, Childs BH, Shi Y, Zinzani PL. Copanlisib plus rituximab versus placebo plus rituximab in patients with relapsed indolent non-Hodgkin lymphoma (CHRONOS-3): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):678-689. doi: 10.1016/S1470-2045(21)00145-5. Epub 2021 Apr 10. PMID 33848462
- [Derived] Morcos PN, Moss J, Veasy J, Hiemeyer F, Childs BH, Garmann D. Model-Based Benefit/Risk Analysis for the Copanlisib Intermittent Dosing Regimen. Clin Pharmacol Ther. 2024 May;115(5):1092-1104. doi: 10.1002/cpt.3173. Epub 2024 Jan 16. PMID 38226495
- See also: Click here to find information about studies related to Bayer AG products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/17067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in North America, South America, South Africa, Europe, Asia, and Australia between 03 August 2015 (first participant first visit) and 15 November 2024 (last participant first visit).
Pre-assignment Details: Overall, 652 were screened and total of 458 participants were randomized in a 2:1 ratio to study treatment: 307 participants to copanlisib/rituximab and 151 participants to placebo/rituximab.
Groups:
- Copanlisib + Rituximab: Copanlisib (60 mg) was administered intravenously (IV) (over approximately 1 h) on Days 1, 8, and 15 of each 28-day cycle. Rituximab (375 mg/m^2) was administered weekly during Cycle 1 on Days 1, 8, 15, and 22, and then on Day 1 of Cycles 3, 5, 7, and 9. Copanlisib was administered before rituximab.
- Placebo + Rituximab: Placebo was administered intravenously (IV) (over approximately 1 h) on Days 1, 8, and 15 of each 28-day cycle. Rituximab (375 mg/m^2) was administered weekly during Cycle 1 on Days 1, 8, 15, and 22, and then on Day 1 of Cycles 3, 5, 7, and 9. Placebo was administered before rituximab.
Period: Overall Study
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Started | 307 | 151
Received Treatment | 304 | 149
Completed (Ongoing with treatment) | 0 | 4
Not Completed | 307 | 147
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Additional primary malignancy | 1 | 1
Not completed — AE not associated with clinical disease progression | 117 | 12
Not completed — AE associated with clinical disease progression | 1 | 4
Not completed — Physician Decision | 2 | 8
Not completed — Non-compliance to study drug | 1 | 0
Not completed — Failure to meet continuation criteria | 1 | 0
Not completed — Switching to other therapy | 2 | 0
Not completed — Withdrawal by Subject | 51 | 16
Not completed — Patient decision: COVID-19 pandemic related | 1 | 0
Not completed — Patient decision | 40 | 14
Not completed — Required procedure failed | 1 | 0
Not completed — Randomized by mistake with study treatment | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive disease - radiological progression | 54 | 80
Not completed — Progressive disease - clinical progression | 6 | 6
Not completed — Drug not administered | 3 | 2
Not completed — Progressive disease | 0 | 1
Not completed — Other reason: Covid-19 pandemic related | 1 | 0
Not completed — Death | 2 | 0
Not completed — Study terminated by sponsor | 19 | 2

BASELINE CHARACTERISTICS:
Population: The number of participants was based on the Full analysis set population and a 2:1 randomization to treatment/placebo groups. Three patients were randomized to the placebo/rituximab arm but received at least one dose of copanlisib by mistake. These patients were included in the copanlisib/rituximab arm in the analysis of safety variables.
Groups:
- Total: Total of all reporting groups
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab | Total
Number analyzed (Participants) | 307 | 151 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (12.1) | 61.5 (11.0) | 61.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 66 | 220
  Male | 153 | 85 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 26 | 55
  Not Hispanic or Latino | 262 | 118 | 380
  Unknown or Not Reported | 16 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 125 | 50 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 164 | 89 | 253
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 7 | 18
Eastern cooperative oncology group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS was measured in a scale from 0 (best) to grade 2, where 0=Fully active, able to carry on all pre-diseases performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2=Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50 percent (%) waking hours (h).
  Participants
    0 - Fully active | 182 | 95 | 277
    1 - Restricted active | 113 | 55 | 168
    2 - Ambulatory and capable of all self-care | 12 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Independent Central Review.
Description: Progression-free survival (PFS) was defined as the time from randomization to progressive disease (PD) or death due to any cause, whichever was earlier according to the Lugano Classification and Response criteria in patients affected by Waldenström macroglobulinemia (kindly refer to the links in the Protocol section).
Time Frame: From first participant randomization (20-Aug-2015) up to data cut-off at primary completion (31-Aug-2020), approximately 5 years and 2-year follow-up after primary completion at 31-Aug-2022, up to 7 years and final analysis at 15-Nov-2024 up to 9 years
Population: All randomized participants (FAS=full analysis set) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months
  At data cut-off=31-Aug-2020 | 21.5 [17.8 to 33.0] | 13.8 [10.2 to 17.5]
  At data cut-off=31-Aug-2022 | 23.2 [19.4 to 33.0] | 13.8 [10.8 to 17.5]
  At data cut-off=15-Nov-2024 | 22.4 [19.7 to 30.7] | 14.0 [11.4 to 19.2]
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — PFS was evaluated with the stratified log-rank test. HR and 95% CI were based on stratified Cox Regression Model; p = 0.000002, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.520, 95% CI 2-sided [0.393 to 0.688]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — PFS was evaluated with the stratified log-rank test. HR and 95% CI were based on stratified Cox Regression Model; p = 0.000003, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.557, 95% CI 2-sided [0.431 to 0.722]
Statistical Analysis 3: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At final analysis; Test type: Superiority — PFS was evaluated with the stratified log-rank test. HR and 95% CI were based on stratified Cox Regression Model; p = 0.000199, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.643, 95% CI 2-sided [0.502 to 0.823]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) was defined as the percentage of participants who have a best response rating over the whole duration of the study (i.e. until time of analysis of PFS) of complete response (CR) or partial response (PR) according to the Lugano Classification and for patients with Waldenström macroglobulinemia (WM) a response rating of CR, very good partial response (VGPR), PR, or minor response (MR) according to the Owen Criteria (kindly refer to the links in the Protocol section).
Time Frame: From first participant randomization (20-Aug-2015) up to data cut-off date at primary completion (31-Aug-2020), approximately 5 years and 2-year follow-up after primary completion at 31-Aug-2022, up to 7 years
Population: All randomized participants (FAS) were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Percentage of participants
  At data cut-off=31-Aug-2020 | 80.8 | 47.7
  At data cut-off=31-Aug-2022 | 80.5 | 49.7
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p < 0.000001, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in ORR = 32.99, 95% CI 2-sided [23.95 to 42.03]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p < 0.000001, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in ORR = 30.67, 95% CI 2-sided [21.63 to 39.72]

3. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate (CRR) was defined as the percentage of participants who had a best response rating over the whole duration of the study (i.e., until the time of analysis of PFS) according to the Lugano Classification and for patients with Waldenström macroglobulinemia (WM) a response rating of Complete Response according to the Owen Criteria (kindly refer to the links in the Protocol section).
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Percentage of participants
  At data cut-off=31-Aug-2020 | 33.9 | 14.6
  At data cut-off=31-Aug-2022 | 34.2 | 15.2
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p < 0.000001, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in CRR = 19.27, 95% CI 2-sided [11.57 to 26.96]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p = 0.000001, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in CRR = 18.92, 95% CI 2-sided [11.11 to 26.73]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as the time (in days) from first observed tumor response Complete Response (CR), Very good partial response (VGPR), Partial Response (PR) or Minor Response (MR) until progression or death from any cause, whichever occurred earlier according to the Owen Criteria (kindly refer to the links in the Protocol section). Only patients with response in FAS were included in the analysis.
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months
  At data cut-off=31-Aug-2020 | 20.4 [17.0 to 30.8] | 17.3 [11.8 to 25.3]
  At data cut-off=31-Aug-2022 | 25.9 [17.7 to 31.5] | 15.2 [12.3 to 25.3]
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — DOR was evaluated with the stratified log-rank test. HR and 95% CI were based on stratified Cox Regression Model; p = 0.030371, Log Rank — 1-sided p-value; Kaplan-Meier estimates = 0.700, 95% CI 2-sided [0.481 to 1.018]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — DOR was evaluated with the stratified log-rank test. HR and 95% CI were based on stratified Cox Regression Model; p = 0.051976, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.761, 95% CI 2-sided [0.547 to 1.059]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was defined as the percentage of participants who had a best response rating as Complete Response (CR), Partial Response (PR) or stable disease (SD) according to the Lugano Classification and for patients with Waldenström macroglobulinemia (WM) as a response rating of CR, very good partial response (VGPR), PR, minor response (MR) or stable disease (SD) according to the Owen Criteria (kindly refer to the links in the Protocol section).
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Percentage of participants
  At data cut-off=31-Aug-2020 | 89.3 | 84.8
  At data cut-off=31-Aug-2022 | 89.3 | 84.8
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p = 0.097339, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in DCR = 4.43, 95% CI 2-sided [-2.26 to 11.12]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — P-value from Cochran-Mantel-Haenszel (CMH) test stratified; p = 0.097339, Cochran-Mantel-Haenszel — 1-sided p-value; Difference in DCR = 4.43, 95% CI 2-sided [-2.26 to 11.12]

6. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time (days) from date of randomization to date of first observed disease progression according to the Lugano Classification and Response criteria in patients affected by Waldenström macroglobulinemia (kindly refer to the links in the Protocol section).
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months
  At data cut-off=31-Aug-2020 | 22.3 [19.4 to 33.2] | 13.8 [10.8 to 18.7]
  At data cut-off=31-Aug-2022 | 27.7 [21.9 to 33.3] | 13.8 [11.0 to 18.7]
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — TTP was evaluated with the stratified log-rank test. HR and 95% CI were based on Cox Regression Model; p < .000001, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.476, 95% CI 2-sided [0.357 to 0.635]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — TTP was evaluated with the stratified log-rank test. HR and 95% CI were based on Cox Regression Model; p < .000001, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.505, 95% CI 2-sided [0.387 to 0.659]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in days) from randomization until death from any cause.
Time Frame: From randomization up to the final analysis at 15-Nov-2024 up to 9 years
Population: All randomized patients (FAS) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months | NA [82.2 to NA] — Value could not be estimated because of censored data (insufficient number of participants with events). | NA [77.3 to NA] — Value could not be estimated because of censored data (insufficient number of participants with events).
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; Test type: Superiority — OS was evaluated with the stratified log-rank test. HR and 95% CI were based on Cox Regression Model; p = 0.436458, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.972, 95% CI 2-sided [0.691 to 1.368]

8. Secondary Outcome: Time to Deterioration in DRS-P (Disease-Related Symptoms - Physical) of at Least Three Points, as Measured by the Functional Assessment of Cancer Therapy Lymphoma Symptom Index-18 (FLymSI-18) Questionnaire.
Description: Time to deterioration in DRS-P (Disease-Related Symptoms - Physical) of at least three points was defined as the time (in days) from randomization to DRS-P decline, progression, or death due to any reason, whichever occurred earlier. The Lymphoma Symptom Index-18 (FLymSI-18) questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and was divided into a total score.
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months
  At data cut-off=31-Aug-2020 | 5.5 [4.2 to 5.9] | 5.5 [4.0 to 7.4]
  At data cut-off=31-Aug-2022 | 5.5 [4.2 to 5.9] | 5.5 [4.1 to 7.4]
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — Time to deterioration in DRS-P was evaluated with the stratified log-rank test. HR and 95% CI were based on Cox Regression Model; p = 0.692610, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 1.060, 95% CI 2-sided [0.843 to 1.331]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.661145, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.841 to 1.302]

9. Secondary Outcome: Time to Improvement in DRS-P (Disease-Related Symptoms - Physical) of at Least 3 Points, as Measured by the Functional Assessment of Cancer Therapy Lymphoma Symptom Index-18 (FLymSI-18) Questionnaire.
Description: Time to improvement in DRS-P (Disease-Related Symptoms - Physical) was defined as the time (in days) from randomization to DRS-P improvement of at least three points. The Lymphoma Symptom Index-18 (FLymSI-18) questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and was divided into a total score.
Time Frame: as for outcome 2
Population: All randomized participants (FAS) were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 151
Months
  At data cut-off=31-Aug-2020 | NA [8.3 to NA] — NA = value cannot be estimated due to censored data (insufficient number of events). | NA [6.0 to NA] — NA = value cannot be estimated due to censored data (insufficient number of events).
  At data cut-off=31-Aug-2022 | 38.5 [8.2 to NA] — NA = value cannot be estimated due to censored data (insufficient number of events). | 35.7 [5.9 to NA] — NA = value cannot be estimated due to censored data (insufficient number of events).
Statistical Analysis 1: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At primary completion date; Test type: Superiority — Time to improvement in DRS-P was evaluated with the stratified log-rank test. HR and 95% CI were based on Cox Regression Model; p = 0.510038, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.996, 95% CI 2-sided [0.732 to 1.355]
Statistical Analysis 2: Comparison: Copanlisib + Rituximab vs Placebo + Rituximab; At 2-year follow-up cut-off date; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.405970, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 1.036, 95% CI 2-sided [0.768 to 1.398]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) at Primary Completion Date.
Description: Adverse events were considered to be treatment-emergent if they have started or worsened after first application of study medication up to 30 days after end of treatment with study medication.
Time Frame: Up to 30 days after end of treatment with study drug, data reporting cut-off at 5 years from the first participant randomization date
Population: Participants in safety analysis set (SAF) with evaluable data reported.
Measure: Number; unit: Participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 146
Participants
  Any TEAEs | 307 | 134
  Any copanlisib- or placebo-related TEAE | 293 | 95
  Any rituximab-related TEAE | 218 | 92

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) at 2-year Follow-up Cut-off Date.
Description: as for outcome 10
Time Frame: Up to 30 days after end of treatment with study drug, data reporting cut-off at 7 years from the first participant randomization date
Population: Participants in safety analysis set (SAF) with evaluable data reported.
Measure: Number; unit: Participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 146
Participants
  Any TEAEs | 307 | 137
  Any copanlisib- or placebo-related TEAE | 295 | 98
  Any rituximab-related TEAE | 218 | 93

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) at Final Analysis
Description: as for outcome 10
Time Frame: Up to 30 days after end of treatment with study drug, data reporting cut-off at final analysis, up to 9 years
Population: Participants in safety analysis set (SAF) with evaluable data reported.
Measure: Number; unit: Participants
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 307 | 146
Participants
  Any TEAEs | 307 | 137
  Any copanlisib- or placebo-related TEAE | 295 | 98
  Any rituximab-related TEAE | 218 | 93

ADVERSE EVENTS:
Time Frame: - Time frame for Serious and Other Adverse Events - from first administration of study drug until 30 days after the last study drug intake. - Time frame for number of death (all causes) - from randomization up to approximately 9 years.
Description: Three patients were randomized to the placebo/rituximab arm but received at least one dose of copanlisib by mistake. These patients were included in the copanlisib/rituximab arm in the analysis of safety variables.
Arm/Group | Copanlisib + Rituximab | Placebo + Rituximab
All-Cause Mortality (participants affected / at risk) | 99/307 | 50/146
Serious Adverse Events (participants affected / at risk) | 161/307 | 32/146
Other Adverse Events (participants affected / at risk) | 298/307 | 127/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib + Rituximab (N=307) | Placebo + Rituximab (N=146)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (7) | 3 (3)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (3)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Eustachian valve hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Administration site extravasation (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Parvovirus B19 infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 22 (25) | 5 (5)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 4 (5) | 2 (3)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 8 (8) | 0 (0)
COVID-19 (Infections and infestations) | 8 (9) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (6) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (27) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (6) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib + Rituximab (N=307) | Placebo + Rituximab (N=146)
Anaemia (Blood and lymphatic system disorders) | 60 (139) | 16 (62)
Neutropenia (Blood and lymphatic system disorders) | 64 (249) | 24 (57)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (32) | 8 (14)
Abdominal pain (Gastrointestinal disorders) | 17 (23) | 6 (7)
Constipation (Gastrointestinal disorders) | 31 (37) | 12 (14)
Diarrhoea (Gastrointestinal disorders) | 106 (245) | 15 (19)
Mouth ulceration (Gastrointestinal disorders) | 21 (31) | 4 (6)
Nausea (Gastrointestinal disorders) | 70 (116) | 17 (25)
Stomatitis (Gastrointestinal disorders) | 41 (59) | 4 (9)
Vomiting (Gastrointestinal disorders) | 45 (62) | 5 (5)
Asthenia (General disorders) | 21 (27) | 5 (7)
Chills (General disorders) | 22 (33) | 7 (10)
Fatigue (General disorders) | 44 (51) | 11 (16)
Influenza like illness (General disorders) | 17 (19) | 7 (10)
Mucosal inflammation (General disorders) | 18 (23) | 2 (2)
Pyrexia (General disorders) | 61 (93) | 14 (21)
Bronchitis (Infections and infestations) | 18 (30) | 8 (9)
Influenza (Infections and infestations) | 8 (9) | 12 (14)
Nasopharyngitis (Infections and infestations) | 28 (41) | 7 (12)
Pneumonia (Infections and infestations) | 36 (54) | 12 (15)
Upper respiratory tract infection (Infections and infestations) | 62 (124) | 28 (37)
Urinary tract infection (Infections and infestations) | 38 (67) | 13 (20)
Oral herpes (Infections and infestations) | 19 (29) | 4 (5)
COVID-19 (Infections and infestations) | 21 (28) | 6 (6)
Alanine aminotransferase increased (Investigations) | 30 (46) | 11 (20)
Amylase increased (Investigations) | 16 (20) | 4 (13)
Aspartate aminotransferase increased (Investigations) | 28 (37) | 12 (22)
Blood bilirubin increased (Investigations) | 16 (31) | 2 (4)
Blood cholesterol increased (Investigations) | 13 (14) | 8 (15)
Blood creatine phosphokinase increased (Investigations) | 25 (41) | 7 (11)
Blood creatinine increased (Investigations) | 16 (26) | 6 (7)
Lipase increased (Investigations) | 18 (39) | 4 (16)
Lymphocyte count decreased (Investigations) | 42 (122) | 9 (38)
Neutrophil count decreased (Investigations) | 102 (434) | 34 (74)
Platelet count decreased (Investigations) | 42 (121) | 12 (23)
Weight decreased (Investigations) | 47 (67) | 4 (5)
White blood cell count decreased (Investigations) | 61 (315) | 17 (53)
Hyperglycaemia (Metabolism and nutrition disorders) | 210 (940) | 35 (93)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 21 (35) | 7 (23)
Hyperuricaemia (Metabolism and nutrition disorders) | 20 (33) | 8 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (38) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 23 (28) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (24) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 13 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (26) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (27) | 5 (6)
Dizziness (Nervous system disorders) | 16 (19) | 6 (6)
Dysgeusia (Nervous system disorders) | 21 (28) | 2 (2)
Headache (Nervous system disorders) | 43 (73) | 10 (20)
Insomnia (Psychiatric disorders) | 18 (19) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (69) | 19 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 14 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (22) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 30 (39) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 35 (51) | 10 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 (33) | 4 (5)
Hypertension (Vascular disorders) | 157 (779) | 31 (119)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT02367040/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02367040/SAP_003.pdf